## The Impact of Mobile Education Delivery on Postoperative Pain Outcomes

Oral Consent Script

IRB Number: 17-04771

NCT number: NA

8/14/2017

## **Oral Consent Script**

Protocol Title: The Impact of Mobile Education Delivery on Postoperative Pain Outcomes

IRB #: 17-004771

Principal Investigator: Amber Stitz

You are being asked to participate in a research study that will evaluate different ways of delivering pain management education and the effect that it has on pain outcomes such as pain scores, participation in treatment, and pain knowledge.

If you agree to participate you will be asked at the start of the study to fill out 2 questionnaire forms one will ask you some demographic and health status questions and the other will assess your knowledge of pain and treatment. These survey's will only take 5 minutes to complete. After surgery, in the hospital, you will receive pain education using either written pamphlets with verbal instruction or an interactive mobile program using an iPad. The type of education you receive will be determined by your location in the hospital after surgery. Before you leave the hospital, you will receive two questionnaires. One will ask you questions about your pain experience while in the hospital. The second survey will assess your knowledge of pain and treatment. This study will not change how your healthcare team will manage your pain after surgery. All study forms will have a unique identifying number so that your information will be kept confidential. Your name and any other identifying information will not be used in the research reports or any related publications. Only your immediate medical records related to this hospital stay and surgery will be accessed by the identified researchers.

If you decide to participate, you will need to read and sign the Authorization to Use and Disclose Protected Health Information (HIPAA) form and return it with the questionnaire. We are not allowed to use the answers without your signature on the HIPAA form. An extra copy is included for your records.

There is minimal risk to you by taking part in this research study. The potential for risk is that the way we deliver the education may meet your needs. If this should happen we will change the education delivery to ensure that you receive all the information the way that best works for you. Additionally, you may feel uncomfortable talking about your pain or other topics included in this study. If you are uncomfortable at any time, you may choose to not answer specific questions or withdraw from study participation.

The benefits which may reasonably be expected to result from this research study are that your overall pain may be lower and you may increase your ability to make informed decisions about your health care and pain treatment options. Other benefits may include less time in the hospital, more satisfaction with your care, and increased self-esteem. However, you may not benefit from participating in this study.

Please understand your participation is voluntary and you have the right to withdraw your consent or discontinue participation at any time without penalty. Specifically, your current or future medical care at the Mayo Clinic will not be jeopardized if you choose not to participate.

If you have any questions about this research study you can contact Amber Stitz at 507-266-3384. If you have any concerns, complaints, or general questions about research or your rights as a participant, please contact the Mayo Institutional Review Board (IRB) to speak to someone independent of the research team at 507-266-4000 or toll free at 866-273-4681.